CLINICAL TRIAL: NCT01448577
Title: A Clinical Records Review Study of the Frequency and Severity of Acute Abdominal "Pancreatitis" Episodes Reported From LPLD Subjects Previously Recruited to Clinical Studies PREPARATION-02, CT-AMT-011-01 and CT-AMT-011-02
Brief Title: Study to Re-assess and Re-confirm Data Previously Recorded About the Incidence and Severity of Acute Abdominal "Pancreatitis" Episodes in Lipoprotein Lipase Deficient (LPLD) Subjects Previously Enrolled on AMT Clinical Studies
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Amsterdam Molecular Therapeutics (Industry)
Collaborators: The Clinical Trial Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CT-AMT-011-03
Record Dates: First submitted 2011-10-03; First posted 2011-10-07 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Lipoprotein Lipase Deficiency
MeSH Terms: conditions — Hyperlipoproteinemia Type I

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dose 3 x 1011 gc/kg: Subjects received AMT-011 at dose 3 x 1011 gc/kg
- Dose 1 x 1012 gc/kg: Subjects received AMT-011 at dose 1 x 1012 gc/kg

SUMMARY:
Lipoprotein lipase deficiency (LPLD) is an autosomal recessive inherited condition caused by homozygosity or compound heterozygosity for mutations within the LPL gene. LPLD results in subjects presenting with fasting plasma triglyceride (TG) levels of > 10 mmol/l. LPLD typically presents in infancy or childhood with usual complaints of severe abdominal pain, repetitive colicky pains and repeated episodes of acute pancreatitis The most severe clinical complication associated with LPLD is acute pancreatitis. Pancreatitis in an LPLD subject often leads to prolonged hospital admissions (sometimes up to weeks). Subjects who survive repeated episodes of acute pancreatitis may develop chronic pancreatitis, ultimately resulting in endocrine and exocrine pancreatic insufficiency.

The clinical manifestations of acute pancreatitis episodes related to LPLD are largely indistinguishable from acute pancreatitis due to other causes. However, collection of data relating to hospital admissions, laboratory test results, scan images and adverse events occurring concomitantly to the acute pancreatic episode should allow elimination of other causes of pancreatitis (e.g gallstones etc) and ultimately allow confirmation of LPLD-related acute pancreatitis. Characterization of the presentation of symptoms which occur around the time of known episodes of LPLD-related acute pancreatitis should also permit identification of episodes of acute pancreatitis which have previously been considered as unrelated or even unrecognized.

The objective of the study is to re-assess and re-confirm data previously recorded about the incidence and severity of acute abdominal "pancreatitis" episodes in LPLD subjects previously enrolled on AMT clinical studies. To assess and document the presentation of acute abdominal episodes that occur around known episodes of pancreatitis and to permit the identification of possible new previously unrecorded episodes of pancreatitis based upon predefined diagnostic criteria. The objective is to recruit the 27 subjects previously enrolled in the above mentioned clinical studies.

DETAILED DESCRIPTION:
Lipoprotein lipase deficiency (LPLD) is an autosomal recessive inherited condition caused by homozygosity or compound heterozygosity for mutations within the LPL gene.

The most severe clinical complication associated with LPLD is acute pancreatitis. Pancreatitis in an LPLD subject often leads to prolonged hospital admissions. Subjects who survive repeated episodes of acute pancreatitis may develop chronic pancreatitis, ultimately resulting in endocrine and exocrine pancreatic insufficiency.

The clinical manifestations of acute pancreatitis episodes related to LPLD are largely indistinguishable from acute pancreatitis due to other causes. However, collection of data relating to hospital admissions, laboratory test results, scan images and adverse events occurring concomitantly to the acute pancreatic episode should allow elimination of other causes of pancreatitis (e.g. gallstones etc) and ultimately allow confirmation of LPLD-related acute pancreatitis. Characterisation of the presentation of symptoms which occur around the time of known episodes of LPLD-related acute pancreatitis should also permit identification of episodes of acute pancreatitis which have previously been considered as unrelated or even unrecognized.

Alipogene tiparvovec (Glybera®) is in development for the therapy of LPLD. In summary, alipogene tiparvovec contains the human lipoprotein (LPL) gene variant LPLS447X in a non-replicating vector in solution administered in a one-time series of intramuscular injections in the arms/legs.

Studies conducted to date with Glybera have evaluated total triglyceride levels as a surrogate marker for efficacy and have not evaluated a clinical endpoint such as acute pancreatitis episodes as a primary endpoint. Post-hoc analysis has suggested that there may be a reduction in the frequency of acute abdominal pancreatitis episodes reported following treatment compared to the frequency reported pre-treatment from past medical history records. The recorded episodes used in this post-hoc analysis were collected from medical history and adverse event data but no uniform criteria were used to classify these as episodes of acute pancreatitis. Review of the post hoc analysis has raised questions that the recorded past medical history of pancreatitis episodes may be inaccurate with respect to diagnosis and number of episodes.

In this case record review study, data will be collected on pancreatitis episodes from subjects who previously enrolled in studies PREPARATION-02 (observational), CT-AMT-011-01 and CT-AMT-011-02. In studies CT-AMT-011-01 and CT-AMT-011-02 subjects received AMT-011 at either dose 3 x 1011 gc/kg or 1 x 1012 gc/kg. Data obtained from medical records, hospital admission/discharge charts, laboratory results and imaging scans will be evaluated for evidence of LPLD-related episodes of pancreatitis by an expert review panel. The evaluation will consider data collected from three time periods:

* subjects entire past medical history,
* the period after enrolment into study but prior to AMT-011 therapy,
* the period post-administration of AMT-011.

Data from the subjects who did not progress to receive AMT-011 will be evaluated as a control group using data collected from past medical history and from the period after enrolment in the PREPARATION-02.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have participated in clinical studies study PREPARATION-02, CT-AMT-011-01 or CT-AMT-011-02,

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who previously enrolled in studies PREPARATION-02 (observational), CT-AMT-011-01 and CT-AMT-011-02
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2010-11; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of acute abdominal "pancreatitis" episodes in LPLD subjects | Retrospective
  To re-assess and re-confirm data previously recorded about the incidence and severity of acute abdominal "pancreatitis" episodes in LPLD subjects previously enrolled on clinical studies PREPARATION-02, CT-AMT-011-02 and CT-AMT-011-02. Acute abdominal episodes will be reviewed and adjudicated using the Atlanta diagnostic criteria for acute pancreatitis

SECONDARY OUTCOMES:
Acute abdominal episodes that occur around known episodes of LPLD pancreatitis | Retrospective
  To assess and document the presentation of acute abdominal episodes that occur around known episodes of LPLD pancreatitis
Previously unrecorded episodes of pancreatitis | Retrospective
  To permit identification as far as possible new previously unrecorded episodes of pancreatitis based upon the Atlanta diagnostic criteria for acute pancreatitis
  * Recorded in LPLD subjects past medical history prior to alipogene tiparvovec therapy, and
  * Recorded in LPLD subjects, post alipogene tiparvovec therapy
Initial onset, duration, and frequency of pancreatitis episodes | Up to 5 years
  To document initial onset, duration, and frequency of pancreatitis episodes in the defined LPLD subject population over a period of five years
Initial onset and presence of chronic pancreatitis | Up to 5 years
  To assess the initial onset and presence of chronic pancreatitis over a period of five years
initial onset and presence of the late complications of chronic pancreatitis | Up to 5 years
  To determine the initial onset and presence of the late complications of chronic pancreatitis including exocrine and endocrine insufficiency over a period of five years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Gaudet, MD, PhD, Principal Investigator — Ecogene-21 Clinical Trial Center Chicoutimi
Locations (2):
- Canada (2):
  - ECOGENE-21 Clinical Trial Center, Chicoutimi, Quebec
  - La Clinique de Maladies Lipidiques de Quebec Inc. (CMLQ, Inc.), Québec, Quebec

REFERENCES:
- [Background] Black DM, Sprecher DL. Dietary treatment and growth of hyperchylomicronemic children severely restricted in dietary fat. Am J Dis Child. 1993 Jan;147(1):60-2. doi: 10.1001/archpedi.1993.02160250062018. PMID 8418601
- [Background] Fortson MR, Freedman SN, Webster PD 3rd. Clinical assessment of hyperlipidemic pancreatitis. Am J Gastroenterol. 1995 Dec;90(12):2134-9. PMID 8540502
- [Background] Santamarina-Fojo S. The familial chylomicronemia syndrome. Endocrinol Metab Clin North Am. 1998 Sep;27(3):551-67, viii. doi: 10.1016/s0889-8529(05)70025-6. PMID 9785052
- [Background] Brunzell JD, Deeb SS. (2001). Familial lipoprotein lipase deficiency, Apo C-ІІ deficiency and hepatic lipase deficiency. In: Scriver CR, Beaudet AL, Sly WS, Valle D, eds. The Metabolic Baisis of Inherited Disease. 8th ED, New York, NY: McGraw-Hill: 2789-2816.
- See also: Sponsor Homepage — http://www.amtbiopharma.com/